CLINICAL TRIAL: NCT05194735
Title: Phase I/II Study of Autologous T Cells Engineered Using the Sleeping Beauty System to Express T-Cell Receptors (TCRs) Reactive Against Cancer-specific Mutations in Subjects With Solid Tumors
Brief Title: Phase I/II Study of Autologous T Cells to Express T-Cell Receptors (TCRs) in Subjects With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCR001-201
Record Dates: First submitted 2021-12-06; First posted 2022-01-18 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Gynecologic Cancer; Colorectal Cancer; Pancreatic Cancer; Non-small Cell Lung Cancer; Cholangiocarcinoma; Ovarian Cancer; Endometrial Cancer; Ovarian Carcinoma; Ovary Neoplasm; Squamous Cell Lung Cancer; Adenocarcinoma of Lung; Adenosquamous Cell Lung Cancer
Keywords: adoptive cell therapy; neoantigen; T cell receptor; T lymphocyte; TCR-engineered T cells; cell therapy; immunotherapy; IL-2; Gene therapy
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Cholangiocarcinoma; Ovarian Neoplasms; Endometrial Neoplasms; Adenocarcinoma of Lung | interventions — aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TCR-T Cell Drug Product (Experimental): Phase I: Dose-escalation of TCR-T Cell Drug Product
  Phase II: Single dose of TCR-T Cell Drug Product after MTD/RP2D determine in Phase I portion of the study
  Interventions: Biological: Neoantigen specific TCR-T cell drug product
- TCR-T Cell Drug Product with Aldesleukin (IL-2) (Experimental): Phase I: Dose-escalation of TCR-T Cell Drug Product with Aldesleukin (IL-2)
  Phase II: Single dose of TCR-T Cell Drug Product with Aldesleukin (IL-2) after MTD/RP2D determine in Phase I portion of the study
  Interventions: Biological: Neoantigen specific TCR-T cell drug product; Biological: Aldesleukin (IL-2)

INTERVENTIONS:
Biological: Neoantigen specific TCR-T cell drug product — Phase I:
  Ascending dose, single Infusion of TCR+ Cells
  Phase II:
  Single infusion at the RP2D
Biological: Aldesleukin (IL-2) — To support growth and activation of TCR-T cell drug product
  Arms: TCR-T Cell Drug Product with Aldesleukin (IL-2)

SUMMARY:
A Phase I/II study of autologous T cells engineered using the Sleeping Beauty transposon/transposase system to express TCR(s) reactive against neoantigens in subjects with relapsed/refractory solid tumors

DETAILED DESCRIPTION:
A Phase I/II study of autologous T cells engineered using the Sleeping Beauty transposon/transposase system to express TCR(s) reactive against neoantigens in subjects with relapsed/refractory solid tumors.

An HLA Typing and Tumor Neoantigen Mutation Testing Protocol (Protocol # TCR001-002) has been used to identify patients for potential enrollment into this Study Protocol. Subjects who have completed the HLA Typing and Tumor Neoantigen Mutation Testing Protocol, i.e., subjects for whom a TCR matching the subject's somatic mutation(s) and HLA type restriction combination is available in Alaunos' TCR library will be eligible for enrollment on this study.

The Phase I part of this study is a prospective, open-label, dose-escalation study of TCR-T cell drug product in patients with progressive or recurrent solid tumors who have failed standard therapy. The Phase II part is a prospective, open-label, single dose portion of the study. The Phase II part will begin once the MTD/RP2D in the Phase I part has been determined.

Subjects with one of the following histologically confirmed solid tumors will be included:

* Cohort 1: Gynecologic cancer (e.g., ovarian, endometrial)
* Cohort 2: Colorectal cancer
* Cohort 3: Pancreatic cancer
* Cohort 4: Non-small cell lung cancer (NSCLC); NSCLC includes but is not limited to squamous cell carcinoma, adenosquamous carcinoma or adenocarcinomas
* Cohort 5: Cholangiocarcinoma

Subject must have a tumor mutation and HLA typing combination that matches to at least one of the following TCRs in the Alaunos' library (mutation & HLA type):

* KRAS G12D & HLA-A*11:01
* KRAS G12D & HLA-C*08:02
* KRAS G12V & HLA-A*11:01
* KRAS G12V & HLA-C*01:02
* TP53 R175H & HLA-A*02:01
* TP53 R175H & HLA-DRB1*13:01
* TP53 R248W & HLA-A*68:01
* TP53 Y220C & HLA-A*02:01
* TP53 Y220C & HLA-DRB3*02:02
* EGFR E746-A750del & HLA-DPA1*02:01, DPB1*01:01

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have completed the HLA Typing and Tumor Neoantigen Identification Protocol (TCR001-002) and for whom a TCR(s) matching the subject's somatic mutation(s) and HLA type restriction combination is available in Alaunos' Clinical TCR library
2. Patients who have previously received at least one line of standard systemic therapy for their advanced/metastatic cancer and have either progressed, recurred, or were intolerant to the previous treatment. Specifically:

   * Subgroup 1. Gynecologic cancers (i.e., ovarian or endometrial):

     1. Ovarian cancer
     2. Endometrial cancer
   * Subgroup 2. Colorectal cancer
   * Subgroup 3. Pancreatic cancer
   * Subgroup 4. Non-small cell lung cancer (NSCLC)
   * Subgroup 5. Cholangiocarcinoma
3. Patients must have evaluable or measurable disease per RECIST 1.1 with at least one lesion that can be measured that is not the biopsied lesion.
4. Patients must be able to provide written informed consent.
5. Patients must be age ≥ 18 years.
6. Clinical Performance Status of ECOG 0 or 1. Approval from the Alaunos Medical Monitor is required for ECOG of 2.
7. Patient must be willing and able to provide written informed consent for the long-term follow-up protocol (TCR001-202) for up to 15 years post TCR-T Cell drug product infusion per FDA requirements.
8. Adequate bone marrow reserves as assessed by the following hematology laboratory criteria:
9. Adequate major organ system function
10. A washout period must have elapsed since completion of any prior systemic therapy, and apheresis with guidelines as follows (windows other than what is listed below should be allowed only after consultation with the Medical Monitor); subjects' non-hematologic toxicities from any prior systemic therapy must have recovered to ≤ Grade 1 (with the exception of neuropathy and alopecia) or baseline prior to starting the protocol's therapy.
11. Patients may have undergone minor surgical procedures or limited-field radiotherapy provided any major organ toxicities have recovered to ≤ Grade 1.
12. Female patients must not be pregnant or breastfeeding.

Exclusion Criteria:

1. Patients with known active CNS metastases
2. Concurrent systemic steroid therapy
3. Any form of primary immunodeficiency
4. Patients who have decreased immune competence
5. History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, aldesleukin or bendamustine
6. Severe chronic respiratory condition
7. History of a bleeding disorder or unexplained major bleeding diathesis
8. Arm B Criteria only: Clinically significant patient history which in the judgment of the principal investigator (PI) would compromise the subject's ability to tolerate high-dose aldesleukin;
9. Any major bronchial occlusion or bleeding not amenable to palliation.
10. Patients with psychiatric illness/social situations at the time of treatment that would limit compliance with study requirements.
11. Participants with known active, uncontrolled bacterial, fungal, or viral infection
12. Patients with a prior history or concurrent malignancy
13. Active unstable or clinically significant medical condition
14. History of any major cardiovascular conditions within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kopetz, MD, PhD, Principal Investigator — MD Anderson
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levy PL, Gros A. Fast track to personalized TCR T cell therapies. Cancer Cell. 2022 May 9;40(5):447-449. doi: 10.1016/j.ccell.2022.04.013. Epub 2022 May 9. PMID 35537408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 participants signed consent forms, 14 participants were apheresed, and 8 participants were lymphodepleted and per the protocol definition were considered enrolled. 8 were treated with TCR-T cells.
Pre-assignment Details: A total of 14 participants underwent apheresis. Per protocol, participants were considered enrolled upon meeting lymphodepletion criteria (n = 8). Six participants were not dosed due to manufacturing failure (n = 2), clinical deterioration (n = 1), or study closure prior to dosing (n = 3). BOIN accelerated dose escalation began with 1 subject at Dose Level 1; additional participants could be enrolled at safe dose levels based on manufactured cell count.
Groups:
- Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells): Participants received a single intravenous infusion of autologous TCR-T cells manufactured at Dose Level 1 (target 5 (1 to <10) × 10⁹ TCR+ cells) following apheresis and manufacturing per protocol. This represents the lowest dose cohort in the sequential dose-escalation design.
- Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells): Participants received a single intravenous infusion of autologous TCR-T cells manufactured at Dose Level 2 (target 40 (10 to <70) × 10⁹ TCR+ cells) following apheresis and manufacturing per protocol. This represents the intermediate dose cohort in the sequential dose-escalation design.
- Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells): Participants received a single intravenous infusion of autologous TCR-T cells manufactured at Dose Level 3 (target 100 (70 to 100) × 10⁹ TCR+ cells) following apheresis and manufacturing per protocol. This represents the highest dose cohort in the sequential dose-escalation design.
Period: Overall Study
Arm/Group | Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells) | Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells) | Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells)
Started | 1 | 13 | 0
Apheresis 1 | 1 | 13 | 0
Apheresis 2 | 0 | 2 | 0
Manufacture 1 | 1 | 12 | 0
Manufacture 2 | 0 | 2 | 0
Lymphodepletion (Enrollment) | 1 | 7 | 0
TCR Infusion | 1 | 7 | 0
Assigned Dose Level 2 But Received Dose Level 1 Due to Manufacturing Process | 0 | 2 | 0
Completed | 1 | 7 | 0
Not Completed | 0 | 6 | 0
Not completed — Apheresed but not administered TCR-T cells due to manufacturing failure | 0 | 1 | 0
Not completed — Apheresed but not administered TCR-T cells due to participant developed brain metastases | 0 | 1 | 0
Not completed — Apheresed but not administered TCR-T cells due to early termination of study | 0 | 3 | 0
Not completed — Cells manufactured but not infused due to participant cerebrovascular accident | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes all participants who were enrolled, apheresed, and received TCR-T cells.
Groups:
- Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells): Participants who received a single infusion of TCR-T cells manufactured at Dose Level 1.
- Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells): Participants who received a single infusion of TCR-T cells manufactured at Dose Level 2.
- Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells): Participants who received a single infusion of TCR-T cells manufactured at Dose Level 3.
- Total: Total of all reporting groups
Arm/Group | Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells) | Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells) | Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells) | Total
Number analyzed (Participants) | 1 | 7 | 0 | 8
Age, Continuous [Median (Full Range); unit: years] | 35 | 54 [50 to 66] |  | 54 [35 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 0 | 5
  Male | 0 | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 |  | 1
  Not Hispanic or Latino | 0 | 7 |  | 7
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 1 | 4 |  | 5
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 2 |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 7 |  | 8
Tumor Type [Count of Participants; unit: Participants]
  Colorectal | 0 | 4 | 0 | 4
  Pancreatic | 0 | 3 | 0 | 3
  Non-small cell lung cancer | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) were defined as any adverse event that began or worsened after initiation of lymphodepletion and up to 28 days following TCR-T cell infusion. TEAEs were coded using MedDRA and summarized by system organ class and preferred term, severity, and relationship to study treatment. Participants were followed for delayed or ongoing toxicities for up to 1 year.
Time Frame: From initiation of lymphodepletion through Day 28 after TCR-T cell infusion, and through long-term follow-up for up to 1 year.
Population: Participants who received a TCR-T cell infusion (Safety Analysis Set).
Measure: Number; unit: participants
Arm/Group | Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells) | Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells) | Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells)
Number analyzed (Participants) | 1 | 7 | 0
participants
  Any TEAE | 1 | 7 |
  Drug-related TEAE | 1 | 7 |
  Drug-related Grade 3 or higher TEAE | 1 | 6 |
  TEAE leading to death | 0 | 0 |
  Treatment-emergent SAE | 1 | 2 |

2. Primary Outcome: Frequency of Dose Limiting Toxicities
Description: Number of participants experiencing DLTs, defined as specific adverse events attributable to the TCR-T cell drug product occurring within the first 28 days of infusion. DLTs include, but are not limited to, Grade 4 neutropenia lasting ≥ 14 days, Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with significant bleeding, and ≥ Grade 3 febrile neutropenia with hemodynamic compromise. Non-hematologic DLTs include Grade 3 or 4 Cytokine Release Syndrome (CRS) that does not improve to Grade ≤ 2 within 72 hours, and Grade 3 Immune-effector cell-associated neurotoxicity syndrome (ICANS) that does not resolve to Grade ≤ 2 within 7 days, among others. The severity of adverse events will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Time Frame: From Day 0 to Day 28 post TCR-T cell drug product infusion.
Population: Participants who received the planned TCR-T cell infusion and either experienced a DLT or completed the 28-day DLT observation period; those with major protocol deviations unrelated to safety during this period were considered non-evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells) | Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells) | Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells)
Number analyzed (Participants) | 1 | 7 | 0
Participants | 0 | 0 |

3. Primary Outcome: Determination of Maximum Tolerated Dose (MTD) or Recommended Phase II Dose (RP2D)
Description: The MTD and/or RP2D was to be determined based on dose-limiting toxicities observed during the dose-escalation phase. The planned definition required ≥2 patients at a given dose level to experience a DLT to declare that dose not tolerated.
Time Frame: From Day 0 to Day 28 post TCR-T cell drug product infusion.
Population: All participants who received a TCR-T infusion and were monitored for DLTs were included in a single analysis population. Eight participants were infused (6 at Dose Level 1, 2 at Dose Level 2). The MTD/RP2D could not be determined because the study closed early before enough evaluable participants were treated to allow formal determination.
Measure: Number; unit: Dose level of TCR-T cells infused
Groups:
- All Dose Levels (DLT-Evaluable Population): Includes all participants who received a TCR-T cell infusion and were monitored for DLTs across all dose levels (6 participants at Dose Level 1 and 2 participants at Dose Level 2; total = 8).
Arm/Group | All Dose Levels (DLT-Evaluable Population)
Number analyzed (Participants) | 8
Dose level of TCR-T cells infused | NA — The MTD or RP2D could not be determined because the study closed early before sufficient participants were treated and evaluated for DLTs to allow formal determination.

4. Secondary Outcome: Feasibility of TCR-T Cell Drug Product Manufacturing
Description: Feasibility will be assessed by the number of participants who met eligibility criteria at each step of the manufacturing process, including inability to undergo apheresis, failure of product manufacture, manufactured product not infused, and successful manufacture and infusion of TCR-T cell drug product.
Time Frame: From apheresis collection to the release of the final TCR-T cell drug product for infusion, estimated to be approximately 5 weeks
Population: The feasibility analysis included 14 participants who underwent apheresis with intent to manufacture TCR-T cell product. Although only 8 met criteria for lymphodepletion and were considered formally enrolled per protocol, all 14 apheresed participants were included for feasibility assessment because manufacturing could be attempted for each.
Measure: Number; unit: participants
Groups:
- Apheresed Participants (Feasibility Population): Includes all 14 participants who underwent apheresis with intent to manufacture TCR-T cell drug product. Although only 8 met criteria for lymphodepletion and were considered enrolled per protocol, all 14 were included for assessment of manufacturing feasibility.
Arm/Group | Apheresed Participants (Feasibility Population)
Number analyzed (Participants) | 14
participants
  Unable to be apheresed for logistical or medical reasons | 0
  Apheresis performed but manufacturing not initiated due to study closure | 2
  Product was successfully manufactured but not administered due to progression or comorbidity. | 2
  Infused successfully at the planned dose after 1 manufacturing round. | 6
  Infused at a lower dose than planned after 1 manufacturing round. | 1
  Infused at a lower dose than planned after 2 manufacturing rounds. | 1
  Patients who were manufacturing failures after 2 manufacturing rounds. | 1
  Product was successfully manufactured but not administered due to study closure. | 1

5. Secondary Outcome: TCR-T Cell Persistence
Description: Persistence of TCR-T cells in peripheral blood was assessed by quantitative PCR for vector copy number per 1 × 10⁶ cells at baseline (1 week prior to infusion), predose (Day 0), and multiple post-infusion time points through Month 18. Only quantifiable values are summarized. Samples with "Not Detected (ND)" or "Below the Limit of Quantitation (BLOQ)" are reported as NA and excluded from summary statistics.
Time Frame: Baseline through Month 18 post-infusion.
Population: Persistence analyses included the 8 participants who received TCR-T infusion (1 at Dose Level 1 and 7 at Dose Level 2). A total of 14 participants underwent apheresis, but only infused participants were evaluable for persistence. Samples with "Not Detected (ND)" or "Below the Limit of Quantitation (BLOQ)" were not quantifiable and are reported as NA. Participants without samples at a given time point were excluded.
Measure: Median (Full Range); unit: copies/1x10^6 cells
Arm/Group | Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells) | Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells) | Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells)
Number analyzed (Participants) | 1 | 7 | 0
copies/1x10^6 cells
  Baseline (1 week prior to infusion) | NA — Values listed as "Not Detected (ND)" or "Below the Limit of Quantitation (BLOQ)" could not be quantified by the qPCR assay and are therefore reported as NA. | NA [0 to 0] — Values listed as "Not Detected (ND)" or "Below the Limit of Quantitation (BLOQ)" could not be quantified by the qPCR assay and are therefore reported as NA. |
  Predose Day 0: number analyzed (Participants) | 1 | 6 | 0
  Predose Day 0 | NA — Values listed as "Not Detected (ND)" or "Below the Limit of Quantitation (BLOQ)" could not be quantified by the qPCR assay and are therefore reported as NA. | NA [0 to 0] — Values listed as "Not Detected (ND)" or "Below the Limit of Quantitation (BLOQ)" could not be quantified by the qPCR assay and are therefore reported as NA. |
  Post Dose Day 0: number analyzed (Participants) | 1 | 6 | 0
  Post Dose Day 0 | 4,240,000 | 2,570,000 [779,000 to 3,970,000] |
  Day 1 | 3,190,000 | 59,200 [20,700 to 1,710,000] |
  Day 2 | 2,640,000 | 408,000 [0 to 2,270,000] |
  Day 4 | 3,500,000 | 570,000 [18,700 to 3,400,000] |
  Day 7 | 743,000 | 101,000 [5,320 to 3,730,000] |
  Day 10 | 674,000 | 112,000 [14,200 to 961,000] |
  Day 14 | 984,000 | 112,000 [7,900 to 938,000] |
  Day 21 | 504,000 | 41,300 [1,140 to 489,000] |
  Day 28 | 404,000 | 32,100 [0 to 297,000] |
  Week 6 | 197,000 | 27,800 [0 to 203,000] |
  Week 12: number analyzed (Participants) | 1 | 5 | 0
  Week 12 | 163,000 | 27,200 [1,960 to 121,000] |
  Month 3: number analyzed (Participants) | 0 | 1 | 0
  Month 3 |  | 42,400 |
  Month 6: number analyzed (Participants) | 1 | 1 | 0
  Month 6 | 88,100 | 8,120 |
  Month 15: number analyzed (Participants) | 0 | 1 | 0
  Month 15 |  | NA — Values listed as "Not Detected (ND)" or "Below the Limit of Quantitation (BLOQ)" could not be quantified by the qPCR assay and are therefore reported as NA. |
  Month 18: number analyzed (Participants) | 0 | 1 | 0
  Month 18 |  | NA — Values listed as "Not Detected (ND)" or "Below the Limit of Quantitation (BLOQ)" could not be quantified by the qPCR assay and are therefore reported as NA. |

6. Secondary Outcome: Percent Change in TCR-T Cell Count From Post Dose to Day 28
Description: Assessed by comparing each participant's highest post-dose TCR-T cell count (copies per 1×10⁶ cells by qPCR) to the TCR-T cell count at Day 28. Percent change was calculated as: ((Day 28 - peak post-dose) / peak post-dose) × 100.
Time Frame: Post-dose through Day 28
Population: 8 participants received TCR-T infusion and were included in the analysis (1 assigned at Dose Level 1, 7 assigned at Dose Level 2).
Measure: Median (Full Range); unit: percent change from peak post dose
Arm/Group | Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells) | Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells) | Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells)
Number analyzed (Participants) | 1 | 7 | 0
percent change from peak post dose | -90.5 | -96.7 [-100 to -91.1] |

ADVERSE EVENTS:
Time Frame: From initiation of lymphodepletion until the participant's final study visit, up to approximately 1 year after TCR-T cell infusion.
Description: Adverse events (AEs) were collected from initiation of lymphodepletion through 28 days after TCR-T cell infusion and during long-term follow-up for up to 1 year. AEs were graded for severity using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 and coded using the Medical Dictionary for Regulatory Activities (MedDRA). Treatment-emergent adverse events (TEAEs) were defined as those that began or worsened after initiation of lymphodepletion.
Arm/Group | Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells) | Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells) | Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells)
All-Cause Mortality (participants affected / at risk) | 1/1 | 6/7 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/7 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 7/7 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells) (N=1) | Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells) (N=7) | Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells) (N=0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 2 (2) | NA
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | NA
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA — Anaemia post chemotherapy
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assigned Dose Level 1 (Target 5 × 10⁹ TCR+ Cells) (N=1) | Assigned Dose Level 2 (Target 40 × 10⁹ TCR+ Cells) (N=7) | Assigned Dose Level 3 (Target 100 × 10⁹ TCR+ Cells) (N=0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 4 (4) | NA
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (5) | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6) | NA
Anaemia (Blood and lymphatic system disorders) | 1 (5) | 7 (36) | NA
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (4) | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | NA
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (5) | NA
Blood fibrinogen increased (Investigations) | 1 (1) | 2 (2) | NA
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
Chills (General disorders) | 1 (1) | 3 (3) | NA
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | NA
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | NA
Cytokine release syndrome (Immune system disorders) | 0 (0) | 3 (4) | NA
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1) | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | NA
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | NA
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Fatigue (General disorders) | 0 (0) | 1 (1) | NA
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (3) | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | NA
Headache (Nervous system disorders) | 1 (1) | 4 (6) | NA
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (6) | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 3 (11) | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 (5) | 2 (3) | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 3 (6) | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | NA
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
Influenza like illness (General disorders) | 0 (0) | 3 (3) | NA
International normalised ratio increased (Investigations) | 1 (1) | 4 (7) | NA
Ketonuria (Renal and urinary disorders) | 0 (0) | 6 (6) | NA
Leukopenia (Blood and lymphatic system disorders) | 1 (9) | 7 (34) | NA
Lymphopenia (Blood and lymphatic system disorders) | 1 (9) | 7 (27) | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
Nausea (Gastrointestinal disorders) | 1 (2) | 5 (6) | NA
Neutropenia (Blood and lymphatic system disorders) | 1 (6) | 7 (41) | NA
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | NA
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | NA
Photophobia (Eye disorders) | 1 (1) | 0 (0) | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Proteinuria (Renal and urinary disorders) | 0 (0) | 3 (5) | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
Pyrexia (General disorders) | 0 (0) | 3 (4) | NA
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (6) | 7 (33) | NA
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
Chest discomfort (General disorders) | 1 (1) | 0 (0) | NA
Clostridium test positive (Investigations) | 0 (0) | 1 (1) | NA
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | NA
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1) | NA
Glycosuria (Renal and urinary disorders) | 0 (0) | 2 (2) | NA
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | NA
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | NA
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | NA
Lipase increased (Investigations) | 0 (0) | 1 (2) | NA
Musculoskeletal pain (General disorders) | 0 (0) | 1 (1) | NA
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
Serum ferritin increased (Investigations) | 1 (1) | 3 (3) | NA
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | NA
Tumour necrosis factor increased (Investigations) | 0 (0) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the clinical trial agreement, the PI may not publish results until after a multi-center publication or a defined period post-study. The sponsor reviews any proposed publication and may delay it to protect proprietary information or file IP. Sponsor controls timing and content of multi-center publications.

DOCUMENTS (2):
  • Study Protocol (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT05194735/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT05194735/SAP_001.pdf